CLINICAL TRIAL: NCT05196126
Title: Comparison of Strategies for Permanent Pacemaker Implantation and/or Cardioneuroablation in Patients With Sinus Node Dysfunction: a Noncommercial Physician-initiated Randomized Controlled Trial
Brief Title: Permanent Pacemaker Implantation or Cardioneuroablation in Sinus Node Dysfunction
Acronym: SANOK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stec, Sebastian, MD, PhD, FESC (Other)
Collaborators: KCRI (Other)
Responsible Party: Principal Investigator, Sebastian Stec, Stec Sebastian MD, PhD, FESC, Stec, Sebastian, MD, PhD, FESC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SANOK
Record Dates: First submitted 2021-10-14; First posted 2022-01-19 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Sinus Node Dysfunction
Keywords: cardioneuroablation; pacemaker; sinus node dysfunction; bradycardia; extracardiac vagal nerve stimulation; ECG monitoring; quality of life
MeSH Terms: conditions — Sick Sinus Syndrome; Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - PACEMAKER (Active Comparator): According with ESC indications for elective pacemaker implantation due to SND will referred for PM implantation.
  Interventions: Procedure: Permament pacemaker implantation
- Group B - CARDIONEUROABLATION (Experimental): According with ESC indications for elective PM implantation due to SND will referred for ICM/ILR implantation or prolonged ECG monitoring. Within 4 weeks patient will be screened by interdisciplinary team and autonomic tests (including atropine tests) will be performed. Than, based on atropine tests, electrophysiologic study and extracardiac vagal nerve stimulation, final indication for cardioneuroablation will be established. Biatrial, binodal cardioneuroablation will be performed with anatomical approach with bilateral extra cardiac vagal nerve stimulation during general anesthesia. Than, patient will be closely monitored and indication for PM implantation will be verified.
  Interventions: Procedure: Cardioneuroablation

INTERVENTIONS:
Procedure: Permament pacemaker implantation — PM implantation
  Arms: Group A - PACEMAKER
Procedure: Cardioneuroablation — Biatrial, binodal CNA procedure with anatomical approach will be performed with pre- and post procedural extracardiac vagal nerve stimulation in general anesthesia.
  Other Names: Extracardiac vagal nerve stimulation
  Arms: Group B - CARDIONEUROABLATION

SUMMARY:
This is a noncommercial, physician-initiated, monitored, multicenter, prospective randomized clinical trial, a proof-of-concept study, investigating a treatment strategy only. The study will use medical products applied for invasive and nonivasive procedures performed at the participating centers.

DETAILED DESCRIPTION:
All patients meeting the inclusion criteria and not meeting the exclusion criteria will be invited to participate in the study. The patient will receive an informed consent form describing the study protocol. After speaking to the investigator and receiving detailed answers to all questions, the patient will sign the written informed consent form to participate in the study or will choose to opt out of randomization and to be included in the registry only.

Premenopausal women who will provide consent to participate in the study will undergo a pregnancy test before any invasive procedure. During the 12-month study duration, the use of effective contraception is recommended.

The patient will be asked to complete the questionnaires on bradycardia symptoms and quality of life (QOL).

Any patient included in the study will be randomized into group A or group B. Patients included in the registry (group C) will undergo patient-tailored interventions and treatments through shared decision-making with a possibility of permanent cardiac pacing (subgroup CA), vagal nerve stimulation (VNS) according to the protocol and cardioneuroablation (subgroup CB), as well as observation (subgroup CO).

ELIGIBILITY:
Inclusion Criteria:

* Age, 18-75 years
* Sinus node dysfunction/disease fulfilling criteria for elective pacemaker implantation according to current ESC guidelines (I, IIa, and IIb )
* Optimization of chronic disease treatment
* Ability to provide informed consent to participate in the study
* Ability to understand patient information.

Exclusion Criteria:

* Contraindications to invasive and noninvasive procedures used in the study
* Uncontrolled endocrine and systemic disorders
* Persistent atrial fibrillation
* Dilated cardiomyopathy
* Severe congenital heart valve disease or cardiomyopathy
* Functional NYHA class III/IV
* Left ventricular ejection fraction <35%
* Left atrial diameter >50 mm
* Previous catheter ablation
* Contraindications to anticoagulant treatment
* Contraindications to catheter ablation
* Chronic, advanced two- or third-degree atrioventricular block associated with structural heart disease
* Contraindications to noninvasive tests
* Pregnancy and lactation
* Previous cardiac surgery
* Implanted pacemaker device
* Neck and chest abnormalities
* Myocardial infarction in the previous 6 months
* Percutaneous coronary intervention in the previous 3 months
* Estimated survival <24 months
* Participation in another drug or medical device program
* Limited capacity to understand the study protocol or psychological disorders precluding informed consent to participate in the study.
* Any other uncontrolled chronic diseases, neck and chest abnormalities, or disorders that constitute a contraindication to catheter ablation, antiarrhytmic treatment, general anesthesia, or extracardiac vagal nerve stimulation (ECANS)
* Severe obesity (body mass index ≥40 kg/m2 )

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Had Freedom From Bradycardia Symptoms at 6 months | 6 months
  Number of participants who had freedom from bradycardia symptoms at 6 months - for all participants - who had CNA versus PM implanation versus no procedure performed. Trial - patient is randomized to standard PM implatantion (Group A) or CNA procedure (Group B). Registry (Group C) - patient refused participation in the trial, and decided to have share-decision making procedure (CNA, PM implanatation) or no intervention at all - taking into account evidence, risk-benefit assesments, expected outcomes and individual patient preferences.
Number of Participants with Pacemaker Implantation at 6 months | 6 monhts
  Number of participants with PM implantation at 6 months

SECONDARY OUTCOMES:
Number of Events of Procedural Complications | 0-6 months
  Procedural Complications (death, stroke, myocardial infarction, heart failure, conduction abnormalities, pericardial effusion requiring drainage, hematoma, pseudoaneurysm (0-6 month changes)
Number of Participants With Post-ablation Inducibility of Sinus Arrest and/or AV Block by Vagal Nerve Stimulation | 1 day (peri-procedural)
  Number of participants with post-ablation inducibility of sinus arrest and/or AV block in pre- and post- procedural extracardiac Vagal Nerve stimulation
Effect of CNA on Quality of Life Parameters Based on EQ-5D-5L Questionnaire | 0, 3, 6, 9, 12 months
  EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on a scale of 1-5 ponts, that describes the patient's health state. The maximum score of 1 indicates the best health state, higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health, 0 indicating the worst health status.
Effect of CNA on Quality of Life Parameters Based on SF-36 Questionnaire | 0, 3, 6, 9, 12 months
  SF-36 questionnaire consists of 36 questions that are distributed across eight scales. Each scale is directly transformed into 0-100 scale. The lower the score the more disability, the higher the score the less disability.
Effect of CNA on Fatigue Based on Modified Fatigue Impact Scale (MFIS) | 0, 6, 12 months
  MFIS is a validated, standardized, 21-item questionnaire, which provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. Total scores range from 0-84. The lower the score the less fatigue, the higher the score the more fatigue impairs physical, cognitive, and psychosocial functioning.
Effect of CNA on Depression/Anxiety based on Modified Hospital Anxiety and Depression Scale (HADS-M) | 0, 6, 12 months
  HADS-M is a validated, standardized 16-item questionnaire to evaluate the association between anxiety and depression and the degree of illness acceptance in patients. Total scores range from 0-64. Higher scores indicate a greater degree of anxiety or depression.
Effect of CNA on Sleep Disorders Based on Epworth Sleep Scale (ESS) | 0, 6, 12 months
  The ESS score is a standardized, validated 8-item questionnaire (with scores 0-3 each). The total score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Effect of CNA on Sleep Disorders Based on Athens Insomnia Scale-8 (AIS-8) | 0, 6, 12 months
  AIS-8 is a standardized, validated questionnaire assessing 8 factors related to nocturnal sleep and daytime dysfunction, which are rated on a 0-3 scale. The sleep is evaluated from the cumulative score of all factors and reported as an individual's sleep outcome. Higher score indicates more sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Stec, MD, PhD, Study Chair — Medical Center SABAMED Medicans
Locations (4):
- Poland (4):
  - Center of Interventional Cardiology, Electrotherapy and Angiology G.V.M. Carint, Ostrowiec Świętokrzyski
  - Medical Center SABAMED, Rzeszów
  - Subcarpatian Center for Cardiovascular Interventions, Laboratory of Electrophysiology, Cardioneuroablation, Ablation, Arrhythmia and Heart Electrostimulation, G.V.M. Carint, Sanok
  - Department of Cardiology, Laboratory of Invasive Electrophysiology, 4th Military Teaching Hospital in Wroclaw, Wroclaw

IPD SHARING:
Plan to Share IPD: No